CLINICAL TRIAL: NCT02063451
Title: Neurohormonal & Behavioral Correlates of Obesity and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Brain Research Foundation (Other)
Responsible Party: Principal Investigator, Amy E Rothberg, Associate Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IWMCNI_01; 5K01DK092322 (NIH)
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Obesity
Keywords: Obesity [C18.654.726.500]; Receptor, Opioid, mu [D12.776.543.750.100.620.550]; Brain [A08.186.211]; Affect [F01.470.047]
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese, Weight Loss, Very Low Calorie Diet (Other): Obese individuals will a Very Low Calorie Diet (VLCD) using the HMR meal replacement (Health Management Resources, Boston, MA) for 3-6 months until individually targeted weight loss determined by a clinician is reached. Typically, individuals consume 850-1000 kilocalories per day.
  Interventions: Dietary Supplement: Very Low Calorie Diet (VLCD)
- Lean, baseline measure (No Intervention): MOR binding will be observed in lean individuals at one timepoint. Lean individuals will not receive any intervention.

INTERVENTIONS:
Dietary Supplement: Very Low Calorie Diet (VLCD) — Very Low Calorie Diet (VLCD) using the HMR meal replacement (Health Management Resources, Boston, MA). Typically, individuals consume 850-1000 kilocalories per day until a targeted 15% reduction in body weight is achieved.
  Arms: Obese, Weight Loss, Very Low Calorie Diet

SUMMARY:
Obesity has reached epidemic levels in the United States, and is on the rise in many industrialized nations. The rate of recidivism for long-term weight loss is substantial and presents a critical problem given the importance of obesity as a modifiable risk factor for diseases like type 2 diabetes. Further, the comorbidity of depression with diseases like obesity, type 2 diabetes, and cardiovascular disease suggest that there may be an underlying shared biology for diseases of metabolic dysfunction and emotional dysregulation. The shared biology of these diseases may actually promote the precipitation and exacerbation of comorbid conditions, impacting the success of treatment. Endogenous opioid systems regulate a number of physiological and psychological processes including mood, energy management, and reward. Endogenous opioid µ-receptor-mediated reward processing is thought to be involved both in the short-term control of eating and hedonic food consumption, based on data in animal models. The present proposal will examine the function of the µ-opioid receptor (MOR) system in lean and obese human volunteers following an overnight fast and the change in µ-opioid receptor occupancy (i.e., endogenous opioid release) following the consumption of a standardized meal using PET imaging with the µ-selective radiotracer [11C]carfentanil. The obese individuals will be retested in the fasting and fed state following a 15% weight loss with a Very Low Calorie Diet. Further, the investigators will evaluate the function of the MOR system within the context of the individual's metabolic and psychological profile including aspects of mood and inhibitory control. This information will provide the neurobiological bases to develop novel avenues of intervention based on individual variations in central mechanisms associated with motivational systems and appetite and their potential role in weight regain.

The investigators hypothesize that overeating in chronically obese individuals will be associated with a dysregulation of MOR system function, manifested by reductions in baseline MOR availability (binding potential, BP) in limbic and reward circuitry, and lower release of endogenous opioids after a standard meal, compared to lean volunteers. The latter is observed as acute reductions in the BP measure after meal ingestion.

DETAILED DESCRIPTION:
Neuroimaging Study. Male and Female volunteers will be recruited from the Investigational Weight Management Clinic (IWMC) at the University of Michigan for this study. All neuropsychological instruments will be collected in lean and obese individuals at baseline, and between 4-6-months. Obese individuals will undergo 4 PET scans: 1) at baseline following an overnight fast; 2) at baseline following consumption of an Ensure shake; 3) after at least a15% reduction in body weight following an overnight fast; 4) and following consumption of an Ensure shake at the post-weight loss time point. Lean individuals will undergo the two scans at baseline after fasting and post-Ensure shake consumption. All lean subjects will consume their normal diets prior to the initial scanning. The obese subjects will undergo their second set of scans, post-weight loss, while still consuming the HMR diet.

Neuroimaging Measures. Two PET studies with [11C]carfentanil (a selective µ-opioid receptor radiotracer) will be acquired for each lean volunteer and 4 PET studies with [11C]carfentanil will be acquired for obese individuals. Structural and functional MRI will be acquired for obese individuals before and after weight loss, and for lean individuals at baseline for co-registration and anatomical standardization of the PET data and activation response to visual stimuli. After their completion, the following data will be used for statistical analyses: 1) Baseline µ-opioid receptor availability in vivo (binding potential, BPND) in lean and obese individuals following an overnight fast. 2) µ-opioid system activation after consuming 500 kcal (16fl oz, 18% protein, 14% CHO, 25% fat) of Ensure shake (fed) in lean and obese individuals as measured by acute reductions in BPND. 3) Baseline MOR BPND in obese individuals who have lost ≥15% of their body weight over 4-6 months (fasting), following an overnight fast. 4) µ-opioid system activation in obese individuals who have lost ≥15% of their body weight after consuming 250 kcal of Ensure shake (fed).

PET Acquisition. Briefly, [11C]carfentanil a selective and specific µ-opioid receptor radioligand, is administered at tracer doses using a bolus/continuous infusion protocol to achieve rapid steady-states between specific and non-specific binding regions (5-7 min post-tracer administration). Twenty-eight frames will be acquired over 70 minutes with an increasing duration (30 sec to 5 min). Two scans will be acquired twice each: A baseline, without challenges, and a scan following consumption of an Ensure shake. Subsequently, dynamic image data for the receptor scans is transformed, on a voxel-by-voxel basis, into parametric maps, and co-registered to each other. These include, 1) a tracer transport measure (K1 ratio, proportional to cerebral blood flow; tracer transport = blood flow x tracer extraction), and receptor-related measures, (BPND), during 2) baseline scans, and 3) following shake consumption. The reduction in BPND from baseline to post-shake consumption represents a measure of endogenous opioid system activation following shake consumption (related to the occupancy and ligand-receptor interactions by the endogenous ligand). These parametric images are calculated using a modified Logan graphical analysis, with the occipital cortex as the reference region. PET images are then co-registered to the T1 MRI structural, anatomical image, affine transformed and warped to standard Montreal Neurological Institute (MNI) stereotactic space using mutual information algorithms. The baseline scan, in the fasted state, will precede the post-consumption scan due to time constraints, and to avoid carry-over effects from active (fed) to baseline (fasted) states. Both PET scans will be performed on the same day to reduce travel time for the subjects and hence experimental burden.

Clinical Measures Psychobehavioral measures to be acquired during the imaging studies include: The Positive and Negative Affect Scale, Profile of Mood Scales, State portion of the Spielberg Anxiety Inventory, and a visual analog scale (VAS) for appetite and palatability will be administered before and after each experiment. These measures will assess emotional state and appetite for correlative purposes with changes in neuroreceptor and circulating hormone levels during performance of the studies. The MINI International Neuropsychiatric Interview (MINI600), Inventory of Depressive Symptomatology (IDS-SR), EuroQol measure of health outcome, Trait portion of the Anxiety Inventory, and NEO Personality Inventory will be obtained prior to scanning for secondary analyses (e.g. relationship between imaging measures and "stable" traits).

ELIGIBILITY:
Inclusion Criteria:

* Obese population defined as BMI > 30 kg/m2.
* Lean population BMI < 28 but > 17 kg/m2.
* Able and willing to provide written informed consent for the trial.
* Right handed
* age >/= 18 years

Exclusion Criteria:

* Evidence of inherited disorders of lipid metabolism.
* History of Cancer within the last 5 years except for minor skin cancers
* Human immunodeficiency virus (HIV) antibody positive.
* Patients with solid organ transplants.
* Positive pregnancy screen in Women
* Uncontrolled thyroid disease
* Unstable angina or NY heart association class II failure or above
* Gastrointestinal disease specifically GI motility disorders
* Unstable neuropsychiatric disease including major depression/anxiety, eating disorder such as bulimia or anorexia
* End stage renal or hepatic disease
* Autoimmune disorders (e.g. SLE)
* Body weight fluctuation of more than 5 kg in the previous 3 months
* Prior bariatric surgery
* A history or current alcohol/substance abuse, or opoid abuse/use and change in smoking habits or cessation in the past 6 months.
* Any medical condition, which in the opinion of the investigator would make the patient unsuitable for recruitment, or could interfere with the patient participating in or completing the protocol.
* Unwilling or unable to consent for the study.
* > 300 lbs (gantry table limit).
* having a waist diameter <53 cm (due to fMRI bore diameter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-01-15 (Actual); Study Completion 2013-01-15 (Actual)

PRIMARY OUTCOMES:
Change in [11C]carfentanil binding in brain in response to feeding prior to weight loss | baseline and 60 minutes following shake consumption
  [11C]carfentanil is a µ-opioid receptor selective radiotracer for PET imaging that will be used to asses the function of the µ-opioid receptor (MOR) system in the brains of lean and obese human volunteers. Measurements of [11C]carfentanil binding will be taken following an overnight fast and following the consumption of a standardized meal to determine the change in µ-opioid receptor occupancy (i.e., endogenous opioid release) in response to feeding.
Change in [11C]carfentanil binding in brain in response to feeding post weight loss | baseline and 60 minutes post shake consumption
  [11C]carfentanil is a µ-opioid receptor selective radiotracer for PET imaging that will be used to asses the function of the µ-opioid receptor (MOR) system in the brains of obese human volunteers following diet-induced weight loss. Measurements of [11C]carfentanil binding will be taken following an overnight fast and following the consumption of a standardized meal to determine the change in µ-opioid receptor occupancy (i.e., endogenous opioid release) in response to feeding. Obese individuals will be retested in the fasting and fed state following a 15% weight loss with a Very Low Calorie Diet which is typically achieved within 6 months.

SECONDARY OUTCOMES:
Change in Hunger scores on a visual analog scale in response to feeding at pre weight-loss | baseline and 120 minutes following shake consumption
  Changes in hunger and craving between the fasted (baseline) and fed state will be measured in lean and obese individuals.
Change in Hunger scores on a visual analog scale in response to feeding post weight-loss | baseline and 120 minutes following shake consumption
  Changes in hunger and craving between the fasted (baseline) and fed state will be measured in lean and obese individuals. Obese individuals will be retested in the fasting and fed state following a 15% weight loss with a Very Low Calorie Diet.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Burghardt, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States